CLINICAL TRIAL: NCT04493814
Title: Study of Association Between Quantity (and Percentage) of Visceral Adipose Tissue and NAFLD-linked Liver Stifness as Mesured by Fibroscan in a Retrospective Cohort of Diabetes Mellitus Patients
Brief Title: Study Visceral Adipose Tissue and Liver Stifness in a Retrospective Cohort of Diabetes Mellitus Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2019PI279
Record Dates: First submitted 2020-07-28; First posted 2020-07-30 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-06

CONDITIONS: NAFLD; Type 2 Diabetes
Keywords: NAFLD; NASH; Insulin resistance; Type 2 diabetes; Visceral Adipose Tissue; DXA; Fibroscan; Vibration-Controlled Transient Elastography; Liver cirrhosis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Diabetes Mellitus, Type 2; Insulin Resistance; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort: All the patients with type 2 diabetes followed at Universitary Hospital of Nancy who had undergone a DEXA and a Fibroscan between 2014 and 2019.

SUMMARY:
Non Alcoholic Fatty Liver Disease (NAFLD) is an emergent disease worldwide, and soon the leading cause of hepatic transplant in the USA. Among this high number of patients, the current challenge is to detect or even predict patients at risk of inflammation (Non Alcoholic or Steatohepatitis or NASH) and end-stage fibrosis, which are the best predictors of liver-related mortality.

Visceral obesity is intimately associated with metabolic disease and adverse health outcomes, such as diabetes, and NAFLD. It has been demonstrated that visceral adipose tissue-linked inflammation was a risk factor of stroke, myocardial infarction, and others metabolic-related complications.

The aim of this study was to evaluate the association of the quantity and percentage of Visceral Adipose Tissue by Dual X-Ray Absorptiometry and liver stiffness by Fibroscan in patients with type 2 diabetes, and other predictors of fibrosis such as FIB-4 and Fibrotest. We retrospectively collected the data of all the diabetic patients who had undergone a DEXA and a Fibroscan between January 1st, 2014 and Decembre 31th, 2019, in the Universitary Hospital of Nancy, France.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* Patients who had undergone a VCTE examen at Universitary Hospital of Nancy between January 1st, 2014 and December 31th, 2019
* - Patients who had undergone a DEXA at Universitary Hospital of Nancy with less than one year of difference with VCTE

Exclusion Criteria:

* Viral, ethylic, drug-linked, genetic, self-immune hepatitis, liver cancer or metatasis ; other causes who could interact with fibroscan or biological markers (thrombocytopenia, undernutrition)
* Type 1 diabetes mellitus
* Weight variation (>5% of body weight) between DEXA mesure and Fibroscan mesure
* Fail of VCTE examination
* High alcohol consumption (>30g/day for men and >20g.day for women)
* Pregnant women
* Other causes of secondary hepatic steatosis (drug-linked, parenteral nutrition, rare diseases...)
* Any other pathology that the investigator would consider not compatible with the research
* Patients in any other research protocol three months before inclusion
* Person referred as in the Public Health code (articles L.1121-5, L.1121-7 and L.1121-8) : pregnant or nursing woman, minor adult, major adult under legal protection, adult unable of giving consent
* Person deprived of their liberty by judicial or administrative decision, person under psychiatric care as described in articles L. 3212-1 and L.3213-1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All the patients with type 2 diabetes, followed and Universitary Hospital of Nancy, France, who had undergone a DEXA and a VCTE examination during their care path, in less than a year apart, between 2014 and 2019.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Estimated)
Dates: Start 2020-07 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Association between quantity of Visceral adipose Tissu and Liver Stiffness | July to September 2020
  Visceral adipose tissu in grams mesured by DEXA, and Liver stiffness in kiloPascal mesured par Vibration-Controlled Transient Elastography

SECONDARY OUTCOMES:
Association between percentage of Visceral adipose Tissu and Liver Stiffness | July to September 2020
  Visceral adipose tissu in percentage on total fat mass mesured by DEXA, and Liver stiffness in kiloPascal mesured par Vibration-Controlled Transient Elastography
Association between quantity of Visceral adipose Tissue and histologic Fibrosis | July to September 2020
  Visceral adipose tissu in grams mesured by DEXA, and histologic fibrosis determined on hepatic biopsy.
Association between percentage of Visceral adipose Tissue and histologic Fibrosis | July to September 2020
  Visceral adipose tissu percentage on total fat mass mesured by DEXA, and histologic fibrosis determined on hepatic biopsy.
Determine the diagnostic performances of quantity of Visceral adipose Tissue for histologic fibrosis diagnosis. | July to September 2020
  Visceral adipose tissu in grams mesured by DEXA, and histologic fibrosis determined on hepatic biopsy.
Determine the diagnostic performances of percentage of Visceral adipose Tissue for histologic fibrosis diagnosis. | July to September 2020
  Visceral adipose tissu percentage on total fat mass mesured by DEXA, and histologic fibrosis determined on hepatic biopsy.
Determine the diagnostic performances of different biologic markers for histologic fibrosis diagnosis. | July to September 2020
  Histologic fibrosis determined on hepatic biopsy.
Build an algorithm with Visceral adipose Tissue mesured and biological markers to predict fibrosis. | July to September 2020
  Prediction algorithm for hepatic fibrosis based on different markers

CONTACTS AND LOCATIONS:
Locations (1):
- GUERCI Bruno, Nancy, France

IPD SHARING:
Plan to Share IPD: Undecided